CLINICAL TRIAL: NCT03195218
Title: Validation of High Resolution Microendoscope in the Screening of Cervical Cancer Precursor Lesions in Brazil (UH3 - Brazil)
Brief Title: HRME in the Screening of Cervical Cancer Precursor Lesions in Brazil (UH3 - Brazil)
Acronym: UH3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: William Marsh Rice University (Other); M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRME-UH3; UH3CA189910 (NIH)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Intraepithelial Neoplasia; Intraepithelial Neoplasm, Cervical; Cervical Cancer; Neoplasm Cervix
Keywords: Cancer prevention; Diagnosis; Microendoscope; High Resolution Microendoscope
MeSH Terms: conditions — Carcinoma in Situ; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Trial with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRME examination (Experimental): HRME will capture images from all areas considered abnormal by VIA (visual inspection with acetic acid) and/or colposcopy. In addition, all four quadrants will be probed with HRME to ensure that any non-acetowhite lesions are also observed
  Interventions: Device: HRME examination

INTERVENTIONS:
Device: HRME examination — HRME will capture images from all areas considered abnormal by VIA and/or colposcopy. In addition, all four quadrants will be probed with HRME to ensure that any non-acetowhite lesions are also observed
  Other Names: Diagnostic tool; Microendoscope

SUMMARY:
STUDY PURPOSES: This study aims to evaluate a high resolution microendoscope (HRME): 1) To assess the sensitivity and specificity of the HRME device in the detection of cervical intraepithelial neoplasia grade 2 (CIN2) or histologically more severe lesion (NIC2+) and cervical intraepithelial neoplasia grade 3 (CIN3) or histologically more severe lesion (NIC3+) in a comprehensive case-by-case basis; 2) Compare the accuracy of the HRME device with acetic acid visualization (VIA) and colposcopy. METHODOLOGY: 1,780 women with abnormal Pap Smears (ASCUS+) or positive high-risk human papillomavirus (HPV) test in the cervix performed in the Barretos Cancer Hospital (HCB, Barretos, Brazil) screening program will be recruited, either at Mobile Prevention Units or Fixed Units, who have been referred for diagnostic investigation with colposcopy. The invitation for women to participate in the study will be made immediately before the medical consultation for colposcopy, in the Prevention Department of Barretos Cancer Hospital. Women who decide to participate in this study will sign an Informed Consent Form after invitation and relevant explanations, which will be provided by the researcher in charge or by a representative with previous training appointed by him for the application of the Form in question. During the colposcopy examination, the HRME device will be used to check the presence of precursor lesions in the cervix. HRME will capture images from all areas considered abnormal by VIA and/or colposcopy. Any abnormal areas detected by VIA and/or colposcopy will undergo a biopsy. If no abnormal area is observed, a cervical microbiopsy will be obtained from an apparently normal area examined using HRME. If during the study a precursor disease or cervical cancer is detected in any woman, an appropriate treatment will be offered by Barretos Cancer Hospital according to an institutional protocol.

DETAILED DESCRIPTION:
STUDY DESIGN:

This is an experimental methodological study with a single-arm, unmasked, unicentric, international diagnostic device.

OUTLINES:

1,780 women with abnormal Pap Smears (ASCUS+) or positive high-risk HPV test in the cervix performed in the Barretos Cancer Hospital (HCB, Barretos, Brazil) screening program will be recruited, either at Mobile Prevention Units or Fixed Units, who have been referred for diagnostic investigation with colposcopy. During the colposcopy examination, the HRME device will be used to check the presence of precursor lesions in the cervix.

PRE-TESTING VERIFICATION:

As this research may include cervical biopsy in women with fertility, for safety reasons, the possibility of pregnancy in this group of women will be verified, since biopsy performed in the cervix of pregnant woman increases the risk of abortion. This verification will be performed by means of clinical history (menstrual delay, signs suggesting pregnancy, contraceptive methods, etc.) and also by means of qualitative research on human chorionic gonadotropin in urine. This test is also known as "rapid pregnancy test" or "pharmacy test", with an extensive list of products sold in Brazil and authorized by "Agencia Nacional de Vigilancia Sanitária" (ANVISA, Brazilian Agency of Health Surveillance). The principle of the test involves a single step immunochromatographic method to detect the hormone. Reaction occurs on a reagent strip, where a small amount of urine is deposited. Test result is provided in approximately 2 minutes. Women who are pregnant (or suspected to be pregnant) will not be included in the study, but will be submitted to diagnostic investigation according to the institutional protocol for pregnant women with changes in the cervix at HCB. These women will receive medical orientation and will be referred to a specialized obstetrical service.

COLLECTION OF CERVICAL CYTOLOGY:

Before the diagnostic examinations are performed, the doctor will collect a new cervical cytology (Papanicolaou), which is part of the routine of the Department of Colposcopy for every woman who has an altered Pap Smear or positive HPV test. These samples will be preserved in an ethanol-based preservative medium (SurePath™ Preservative Fluid, Becton & Dickinson, USA) and will be sent to the Department of Pathology of HCB where they will undergo an automated processing for the preparation of cytology slides.

DIAGNOSTIC EXAMINATIONS:

VIA will be performed using 3-5% acetic acid, applied on the cervix and to any abnormal lesions observed. Then, iodine solution will be applied, and the colposcopy will be performed. It is necessary to clarify that the application of acetic acid and iodine is routinely performed during a standard colposcopy examination.

Then, Proflavine (0.01%) will be applied to the surface of the cervix. HRME will capture images from all areas considered abnormal by VIA and/or colposcopy. In addition, all four quadrants will be probed with HRME to ensure that any non-acetowhite lesions are also observed. The person responsible for the colposcopy will take note of your opinion about the lesion and HRME image at each area (normal, benign, low-grade precancerous, high-grade precancerous or cancer). The complete HRME imaging procedure will add 5-10 minutes to the standard colposcopy examination. Observations related to VIA, colposcopy and HRME will be registered by quadrant. Any abnormal areas detected by VIA and/or colposcopy will undergo a biopsy. If no abnormal area is observed, but the woman has an altered cytology test or a positive HPV test, a cervical microbiopsy will be obtained from an apparently normal area captured by HRME imaging of that area. For all cervical biopsies, special tweezers will be used, causing minimal tissue trauma (microbiopsy) and reducing participant discomfort. These tweezers are different from those commonly used in colposcopy tests, which usually perform biopsies on large areas and bring more discomfort to women.

Two experienced HCB pathologists, ignoring all study results, will review histology and classify areas as normal, cervical intraepithelial neoplasia grade 1 (CIN 1), CIN 2, CIN 3, adenocarcinoma in situ (AIS) or cancer according to standardized criteria. Conflicting results will be resolved by means of consensus review among pathologists.

HIGH-RISK HPV SCREENING AND GENOTYPING:

High-risk HPV screening will be performed on aliquots of cervical cytology samples (SurePath™) collected just prior to colposcopy in women who have not been submitted to this test yet. HPV test will be performed on a Cobas X480 ™ device (Roche Molecular Systems, USA), which is available at the technology park of the Molecular Oncology Research Center of Barretos Cancer Hospital - Pio XII Institution. The test protocol will be performed as described by the manufacturer.

COBAS system is an automated amplification device (by means of real time polymerase chain reaction (PCR)) for the detection of 14 high-risk HPV types (16, 18 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68), and can process up to 94 simultaneous samples. Tests which detected high-risk non-16 and non-18 HPV will be submitted to complementary analysis to identify genotype(s) using the linear array technique, since COBAS system does not provide genotyping of these high-risk HPVs. For this purpose, linear array HPV genotyping (CE-IVD) Test for HPV Genotyping kit (Roche Molecular Systems, USA) will be used.

DATA ANALYSIS:

The primary endpoint is the diagnosis rate of CIN2+ and CIN3+. Sensitivity and diagnostic specificity of VIA, colposcopy and HRME based on each lesion and each patient using histological diagnosis as gold standard will be calculated assuming lesions diagnosed as CIN2 + or CIN3 + are positive. Sensitivity and specificity of VIA and colposcopy will also be calculated as a comparison method.

A case-by-case description will be made using descriptive statistics. Categorical variables will be compared by means of the chi-square test or Fisher's exact test, depending on the expected values in the contingency tables. To compare numerical variables, the t-tests or the Mann-Whitney test will be used depending on the adherence to normality (to be verified by the Kolmogorov-Smirnov test).

SAMPLE SIZE CALCULATION:

Sample calculation was based on information from other studies of the same group (including data not yet published). The following premises were taken: HRME sensitivity and specificity for CIN2+ diagnosis (93% and 48%, respectively, per biopsy area) and prevalence of CIN2+ in the colposcopy clinic of HCB (ranging from 20 to 30%). Considering a prevalence of disease of 25% , it is estimated that it will be necessary to include 1,424 women (625 cases for sensitivity calculation and 799 cases for specificity calculation) to reach the expected sensitivity and specificity rates with a maximum margin of error of 4% for a 95% confidence interval. Considering an estimated loss of 10-15% (non-attendance for colposcopy examination and HRME), the corrected sample estimate will range from 1,566 to 1,637 women. Therefore, the study intends to include 1,600 women with abnormal cervical cytology or positive HPV test. Additionally, a group of women with no change in cervical cytology and HPV test will be invited to participate in the research in order to check verification bias. This bias occurs when only the positive cases in the screening are selected to perform complementary diagnostic examinations, overestimating the sensitivity and underestimating the specificity. It is recommended that a percentage of negative cases be verified according to the standard gold examination. Therefore, 10% of the study population will consist of negative cases in both cervical cytology and the HPV test, which corresponds to nearly 180 cases. Thus, the final sample estimate will be of 1,780 women, of whom 1,600 women will have screening (altered cytology or positive HPV test) results reported as positive and 180 will have screening results reported as negative (negative cytology and HPV test).

STUDY SCHEDULE:

The study will last 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and older;
2. Women with abnormal cervical cytology (atypical squamous cells of undetermined significance or more severe interpretations [≥ASC-US]) or positive high-risk HPV test on cervical samples. Additionally, 10% of the study population will consist of women with no change in cervical cytology and HPV test in order to check verification bias (see further explanations in "6.2. Sample calculation");
3. Women with intact cervix or previously submitted to LEEP (loop electrosurgical excision procedure), cone or cryotherapy, with the presence of the cervix;
4. Women of childbearing potential should have a negative urine or blood pregnancy test;
5. Ability to understand and willing to provide informed consent document.

Exclusion Criteria:

1. Women under 18 years old;
2. Women who have undergone hysterectomy with removal of the cervix;
3. Women with known allergy to proflavine or acriflavine;
4. Women who are pregnant or nursing at the time of enrollment;
5. Incapacitated women or in vulnerable situations or who are not willing to give consent;
6. Women who belong to the indigenous community.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1780 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Isolated accuracy of HRME | Biopsy of uterine cervix will be performed during HRME / colposcopy examination
  Sensitivity and Specificity of CIN2+ and CIN3+ detection using HRME

SECONDARY OUTCOMES:
Comparison of accuracy | Biopsy of uterine cervix will be performed during HRME / colposcopy examination
  Comparison of sensitivity and specificity of CIN2+ and CIN3+ with colposcopy and VIA

CONTACTS AND LOCATIONS:
Overall Officials: Rui M Reis, PhD, Study Director — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
RedCap Platform will be used to share data.